CLINICAL TRIAL: NCT05523011
Title: A Phase 1, Open-label Study to Determine Safety and Tolerability of the Topical Application of Mesenchymal Stem/Stromal Cell (MSC) Exosome Ointment to Treat Psoriasis in Healthy Volunteers
Brief Title: Safety and Tolerability Study of MSC Exosome Ointment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paracrine Therapeutics Dermatology Pte. Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTD2021P001
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Psoriasis
Keywords: Mesenchymal stem/stromal cell; Exosome; Exosome ointment; Topical application; Safety and Tolerability; Extracellular vesicle
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Single-center, single-arm, open-label study
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosome Ointment (Experimental): The subjects will apply exosome ointment along with Vesiderm liposome cream (TID per day, 20 days). Each day (from Day 1 to 20), the study product will be applied with a gap of 4 hours between three doses to a healthy area (one hand area) on the forearm using 1 fingertip unit (FTU). The Vesiderm liposome cream is meant to keep the application site moisturized.
  Interventions: Drug: Exosome ointment

INTERVENTIONS:
Drug: Exosome ointment — 100 µg MSC exosomes/g ointment

SUMMARY:
This phase 1 study aims to evaluate the safety and tolerability of the application of the MSC exosome ointment with repeated topical application on adult healthy subjects (TID from Day 1 to 20). The results of this study were to provide the first clinical information on the drug's safety and inform the selection of administration of exosome ointment to be evaluated in subsequent clinical studies. The endpoints included to assess the safety and tolerability of exosome ointment for topical application in healthy adult volunteers are:

* Frequency of treatment-emergent adverse events (TEAEs)
* The incidence rate of local skin responses (LSR, i.e., erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, erosion/ulceration, hyperpigmentation, hypopigmentation, and scarring) [Time Frame: Days 1 and 21]
* Changes from baseline in blood parameters (including hematology, chemistry, and other inflammation parameters such as C-reactive protein [CRP] and erythrocyte sedimentation rate [ESR]) [Time Frame: Days 1 and 21]

DETAILED DESCRIPTION:
This study was conducted in accordance with the protocol and consensus ethical principles derived from international guidelines including the Declaration of Helsinki, Council for International Organizations of Medical Sciences (CIOMS) International Ethical Guidelines, applicable International Conference on Harmonization (ICH), Good Clinical Practice (GCP) Guidelines, and other applicable laws and regulations.

This was a Phase 1, single-center, open-label study. After signing an ICF, subjects underwent screening procedures on Day 1 prior to the first study product application to determine eligibility. Once eligible, all subjects (n=10) received topical treatment with the MSC exosome ointment immediately followed by Vesiderm liposome cream TID on the forearm with a gap of 4 hours between doses.

The study consisted of the following periods:

* A Screening Period of 1 day (Day 1)
* A Treatment Period of 20 days (Day 1 to 20)
* An End of Study (EOS) Period of 1 day (Day 21 [+3 days]).

Screening Period

The subjects were screened for eligibility on Day 1 prior to the application of the study product. Subjects were asked to sign the ICF after having the study described to them. After obtaining written informed consent, subjects underwent the following screening procedures for participation in the study:

* Inclusion/exclusion criteria assessments
* Vital signs
* Medical history
* Demographic data review
* Standard hematology panel
* Renal panel
* Liver function test
* Inflammatory blood examinations
* Pregnancy test (if applicable)
* Concomitant medications

Identification, visual assessment, and photography of application area

A trained expert evaluator (an Investigator or designee) identified the area of study product application and performed visual assessments which were carried out using an adapted version of SCORing Atopic Dermatitis (SCORAD) scale and visual assessment score (VAS). A photograph of the area of application was also taken using a dedicated compact digital camera at the clinic where subject visits were done.

Treatment Period

After confirmation of the application site, the subjects applied exosome ointment along with Vesiderm liposome cream (TID per day). Each day (from Day 1 to 20), the study product was applied with a gap of 4 hours between each dose to a healthy area (one hand area) on the forearm using 1 fingertip unit (FTU). The Vesiderm liposome cream was meant to keep the application site moisturized.

All through the treatment period, the subjects completed the Subject Diary to capture adverse events (AEs; skin-related and other), concomitant medications, and time of study product application.

The site coordinator called the subjects every 3 days (Days 3, 6, 9, 12, 15, and 18) to follow up on the investigational product's (IP) compliance, and if subjects had any adverse events or had taken any concomitant medications during the period. Any AEs reported by the subject during the calls were to be referred to the investigator for appropriate review and follow-up.

End of Study (EOS) Period

The EOS period was on Day 21 (+3 days). The subjects visited the clinic on this day for the assessments such as vital signs, blood examinations (hematology, chemistry, and inflammatory blood examinations), photographs of the area of application, visual assessment of the area of application, AEs, and concomitant medications used.

The assessments at this visit were also to be conducted in case of early termination or withdrawal of any subject.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF prior to entering the study or undergoing any study procedures.
2. Male or female, >21 years of age at the time of signing the informed consent.
3. Subject who had been fully vaccinated for COVID-19 and was not under quarantine or Stay Home Notice or on medical leave.
4. Subject who was willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Subject was able to read and write in the English language.
6. For women who were not postmenopausal (> 12 months of non-therapy induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus):

   1. had a negative pregnancy test at screening
   2. remained abstinent or used contraceptive methods during the treatment period and continued for at least 30 days (one menstrual cycle) after the last treatment dose.

Exclusion Criteria:

1. Subject had any serious skin condition that was not well controlled.
2. Subject was currently using topical treatments.
3. Pregnant or breast-feeding women.
4. Subject had received phototherapy, oral corticosteroids, oral retinoid, oral immunosuppressive / immune modulative drugs, cytostatic / cytotoxic drugs, cyclosporine, or methotrexate within 30 days prior to the first application of the study product.
5. Subject was currently using any medications including biologics or undergoing treatment known to affect skin conditions.
6. Subject had any other clinically significant laboratory abnormalities, co-morbidities or psychiatric conditions that would place the subject at increased risk or confound the objectives of the study.
7. Subject had used any investigational drugs or biologics and/or participated in any clinical trial within the last 60 days before the day of the first dose of the study drug or was taking part in a non-medication study that would interfere with study compliance or outcome assessments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Suyien Chandran, Dr., Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is on a case-by-case basis.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exosome Ointment
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 10
Hematology-Basophils [Mean (Standard Deviation); unit: 10^9 Basophils/L] — number of cell per liter of blood
  10^9 Basophils/L | 0.036 (0.0171)
Hematology-Eosinophils [Mean (Standard Deviation); unit: 10^9 Eosinophils/L] — number of cell per liter of blood
  10^9 Eosinophils/L | 0.144 (0.1121)
Hematology-Hematocrit [Mean (Standard Deviation); unit: %] | 41.56 (5.214)
Hematology-Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.56 (1.896)
Hematology-Lymphocytes [Mean (Standard Deviation); unit: 10^9 Lymphocytes/L] | 1.635 (0.3346)
Hematology-Monocytes [Mean (Standard Deviation); unit: 10^9 Monocytes/L] | 0.371 (0.1381)
Hematology-Red Blood Cell [Mean (Standard Deviation); unit: 10^12 Red blood cells/L] | 4.847 (0.6072)
Hematology-White Blood Cell [Mean (Standard Deviation); unit: 10^9 White blood cells/L] | 5.692 (1.7182)
Renal Panel-Bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 26.4 (1.51)
Renal Panel-Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 10.354 (3.8044)
Renal Panel-Calcium [Mean (Standard Deviation); unit: mmol/L] | 2.290 (0.0887)
Renal Panel-Chloride [Mean (Standard Deviation); unit: mmol/L] | 105.1 (1.66)
Renal Panel-Creatinine [Mean (Standard Deviation); unit: umol/L] | 65.3 (10.92)
Renal Panel-Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.02 (1.094)
Renal Panel-Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.17 (0.445)
Renal Panel-Sodium [Mean (Standard Deviation); unit: mmol/L] | 140.0 (1.56)
Liver Function Test-Alanine transaminase [Mean (Standard Deviation); unit: U/L] | 22.1 (13.56)
Liver Function Test-Albumin [Mean (Standard Deviation); unit: g/L] | 43.0 (2.21)
Liver Function Test-Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] | 64.2 (17.33)
Liver Function Test-Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 20.6 (5.64)
Liver Function Test-Direct bilirubin [Mean (Standard Deviation); unit: umol/L] | 4.3 (2.67)
Liver Function Test-Total bilirubin [Mean (Standard Deviation); unit: umol/L] | 13.0 (9.81)
Inflammatory Blood Examinations-C-reactive protein [Mean (Standard Deviation); unit: mg/L] | 1.88 (2.107)
Inflammatory Blood Examinations-Erythrocyte sedimentation rate [Mean (Standard Deviation); unit: mm/hr] | 13.5 (11.82)
Vital Signs-Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 123.5 (13.72)
Vital Signs-Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79.4 (13.54)
Vital Signs-Heart Rate [Mean (Standard Deviation); unit: beats/min] | 78 (9.85)
Vital Signs-Respiratory Rate [Mean (Standard Deviation); unit: breaths/min] | 16.2 (2.66)
Vital Signs-Body Temperature [Mean (Standard Deviation); unit: degree Celcius] | 36.64 (0.241)
SCORAD-Dryness [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
SCORAD-Oozing/Crusting [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
SCORAD-Redness [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
SCORAD-Scratch marks [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
SCORAD-Skin thickening [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
SCORAD-Swelling [Count of Participants; unit: Participants]
  0(None) | 10
  1(Mild) | 0
  2(Moderate) | 0
  3(Severe) | 0
VAS-Itch [Mean (Standard Deviation); unit: units on a scale] — 0 (no itch) to 10 (worst imaginable itch)
  units on a scale | 0.0 (0.00)
VAS-Sleeplessness [Mean (Standard Deviation); unit: units on a scale] — 0 (no sleeplessness) to 10 (worst imaginable sleeplessness)
  units on a scale | 0.0 (0.00)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: All through the treatment period, the subjects completed the Subject Diary to capture the frequency of TEAEs.
Time Frame: Day 1 - 20
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants | 0

2. Primary Outcome: Change From Baseline in the Systolic Blood Pressure After 20 Days of Treatment
Description: Systolic blood pressure (mmhg) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmHg | -4.3 (10.93)

3. Primary Outcome: Change From Baseline in the Diastolic Blood Pressure After 20 Days of Treatment
Description: Diastolic blood pressure (mmhg) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmHg | -9.4 (12.12)

4. Primary Outcome: Change From Baseline in the Heart Rate After 20 Days of Treatment
Description: Heart rate (beats/min) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
beats/min | 2.3 (10.83)

5. Primary Outcome: Change From Baseline in the Respiratory Rate After 20 Days of Treatment
Description: Respiratory rate (breaths/min) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
breaths/min | 0.5 (3.57)

6. Primary Outcome: Change From Baseline in the Body Temperature After 20 Days of Treatment
Description: Body temperature (°C) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: degree Celcius
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
degree Celcius | -0.07 (0.263)

7. Primary Outcome: Change From Baseline in the Basophils After 20 Days of Treatment
Description: Basophils (10^9 Basophils /L) were assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^9 Basophils /L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^9 Basophils /L | 0.010 (0.0133)

8. Primary Outcome: Change From Baseline in the Eosinophils After 20 Days of Treatment
Description: Eosinophils (10^9 Eosinophils/L) were assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^9 Eosinophils/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^9 Eosinophils/L | 0.005 (0.0276)

9. Primary Outcome: Change From Baseline in the Hematocrit After 20 Days of Treatment
Description: hematocrit(%) assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
percentage change from baseline | 0.44 (0.914)

10. Primary Outcome: Change From Baseline in the Hemoglobin After 20 Days of Treatment
Description: Hemoglobin (g/dL) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
g/dL | 0.13 (0.330)

11. Primary Outcome: Change From Baseline in the Lymphocytes After 20 Days of Treatment
Description: Lymphocytes (10^9 Lymphocytes/L) were assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^9 Lymphocytes/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^9 Lymphocytes/L | 0.059 (0.3152)

12. Primary Outcome: Change From Baseline in the Monocytes After 20 Days of Treatment
Description: Monocytes (10^9 Monocytes/L) were assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^9 Monocytes/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^9 Monocytes/L | -0.004 (0.0936)

13. Primary Outcome: Change From Baseline in the Red Blood Cell After 20 Days of Treatment
Description: Red blood cell (10^12 Red blood cells/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^12 Red blood cells/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^12 Red blood cells/L | 0.034 (0.1101)

14. Primary Outcome: Change From Baseline in the White Blood Cell After 20 Days of Treatment
Description: White Blood Cell (10^9 White blood cells/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: 10^9 White blood cells/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
10^9 White blood cells/L | 0.008 (0.8306)

15. Primary Outcome: Change From Baseline in the Bicarbonate After 20 Days of Treatment
Description: Bicarbonate (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | -1.4 (2.27)

16. Primary Outcome: Change From Baseline in the Blood Urea Nitrogen After 20 Days of Treatment
Description: Blood urea nitrogen (mg/dL) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mg/dL | 1.800 (3.1564)

17. Primary Outcome: Change From Baseline in the Calcium After 20 Days of Treatment
Description: Calcium (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | 0.016 (0.0538)

18. Primary Outcome: Change From Baseline in the Chloride After 20 Days of Treatment
Description: Chloride (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | 0.8 (1.93)

19. Primary Outcome: Change From Baseline in the Creatinine After 20 Days of Treatment
Description: Creatinine (umol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
umol/L | 1.3 (5.66)

20. Primary Outcome: Change From Baseline in the Glucose After 20 Days of Treatment
Description: Glucose (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | -0.19 (1.309)

21. Primary Outcome: Change From Baseline in the Potassium After 20 Days of Treatment
Description: Potassium (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | 0.17 (0.263)

22. Primary Outcome: Change From Baseline in the Sodium After 20 Days of Treatment
Description: Sodium (mmol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mmol/L | 0.4 (1.78)

23. Primary Outcome: Change From Baseline in the Alanine Transaminase After 20 Days of Treatment
Description: Alanine transaminase (U/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
U/L | 0.6 (8.85)

24. Primary Outcome: Change From Baseline in the Albumin After 20 Days of Treatment
Description: Albumin (g/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
g/L | 0.4 (1.90)

25. Primary Outcome: Change From Baseline in the Alkaline Phosphatase After 20 Days of Treatment
Description: Alkaline phosphatase (U/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
U/L | 2.9 (3.11)

26. Primary Outcome: Change From Baseline in the Aspartate Aminotransferase After 20 Days of Treatment
Description: Aspartate aminotransferase (U/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
U/L | 1.3 (5.48)

27. Primary Outcome: Change From Baseline in the Direct Bilirubin After 20 Days of Treatment
Description: Direct bilirubin (umol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
umol/L | 1.0 (1.41)

28. Primary Outcome: Change From Baseline in the Total Bilirubin After 20 Days of Treatment
Description: Total bilirubin (umol/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
umol/L | 1.0 (4.27)

29. Primary Outcome: Change From Baseline in the C-reactive Protein After 20 Days of Treatment
Description: C-reactive protein (mg/L) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mg/L | -0.11 (0.409)

30. Primary Outcome: Change From Baseline in the Erythrocyte Sedimentation Rate After 20 Days of Treatment
Description: Erythrocyte sedimentation rate (mm/hr) was assessed on Day 1 (pre-treatment) and Day 21 (+3 days)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
mm/hr | -2.0 (4.90)

31. Primary Outcome: Assessment of the Dryness of the Area of Application
Description: Visual assessments of the dryness of the area of application was carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
  SCORAD scale assessment (range: 0-3) 0= none, 1= mild, 2= moderate, 3= severe
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

32. Primary Outcome: Assessment of the Oozing/Crusting of the Area of Application
Description: Visual assessments of the oozing/crusting of the area of application was carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
  SCORAD scale assessment (range: 0-3) 0= none, 1= mild, 2= moderate, 3= severe
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

33. Primary Outcome: Assessment of the Redness of the Area of Application
Description: Visual assessments of the rednessof the area of application was carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
  SCORAD scale assessment (range: 0-3) 0= none, 1= mild, 2= moderate, 3= severe
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

34. Primary Outcome: Assessment of the Scratch Marks of the Area of Application
Description: Visual assessments of the scratch marks the area of application were carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
  SCORAD scale assessment (range: 0-3) 0= none, 1= mild, 2= moderate, 3= severe
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

35. Primary Outcome: Assessment of the Skin Thickening of the Area of Application
Description: Visual assessments of the skin thickening the area of application was carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
  SCORAD scale assessment (range: 0-3) 0= none, 1= mild, 2= moderate, 3= severe
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

36. Primary Outcome: Assessment of the Swelling of the Area of Application
Description: Visual assessments of the swelling of the area of application was carried out using an adapted version of SCORAD scale on Day 1 (pre-treatment) and Day 21 (+3 days).
Time Frame: Day 1 - 21+3
Measure: Count of Participants; unit: Participants
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
Participants
  Day 1: 0(None) | 10
  Day 1: 1(Mild) | 0
  Day 1: 2(Moderate) | 0
  Day 1: 3(Severe) | 0
  Day 21+3: 0(None) | 10
  Day 21+3: 1(Mild) | 0
  Day 21+3: 2(Moderate) | 0
  Day 21+3: 3(Severe) | 0

37. Primary Outcome: Assessment of the Itch of the Area of Application
Description: Subjective symptoms: The identified area of application was assessed for the subjective symptom itch, graded from 0 (no itch) to 10 (worst imaginable itch)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
score on a scale
  Day 1 | 0.0 (0.00)
  Day 21+3 | 0.0 (0.00)

38. Primary Outcome: Assessment of the Sleeplessness
Description: Subjective symptoms: The participant was assessed for the subjective symptom sleeplessness and graded from 0 (no sleeplessness) to 10 (worst imaginable sleeplessness)
Time Frame: Day 1 - 21+3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exosome Ointment
Number analyzed (Participants) | 10
score on a scale
  Day 1 | 0.0 (0.00)
  Day 21+3 | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: Treatment period (Day1-Day20)
Description: All through the treatment period, the subjects completed the Subject Diary to capture the frequency of adverse event
Arm/Group | Exosome Ointment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT05523011/Prot_SAP_000.pdf